CLINICAL TRIAL: NCT03507868
Title: Effect of Non-Surgical Periodontal Therapy on Salivary and Gingival Crevicular Fluid YKL-40 and IL-6 Levels in Chronic Periodontitis
Brief Title: YKL-40 and IL-6 Levels in Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Zeynep Pinar KELES (Other)
Responsible Party: Sponsor-Investigator, Zeynep Pinar KELES, ZEYNEP PINAR KELEŞ, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Other Study IDs: 2016/1003
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva and gingival crevicular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Periodontally healthy individuals
- Group 2: Chronic periodontitis patients
  Interventions: Procedure: Nonsurgical periodontal therapy

INTERVENTIONS:
Procedure: Nonsurgical periodontal therapy — Nonsurgical periodontal therapy includes oral hygiene education and scaling and root planning approaches to eliminate microbial dental plaque that is the primary etiology of periodontal diseases.
  Groups: Group 2

SUMMARY:
The primer aim of the study was to investigate saliva and gingival crevicular fluid (GCF) YKL-40 and also interleukin-6 (IL-6) levels in chronic periodontitis pathogenesis.

DETAILED DESCRIPTION:
This study consisted of two groups: 26 periodontally healthy individuals and 26 generalized chronic periodontitis patients. Chronic periodontitis patients were received nonsurgical periodontal treatment. Clinical measurements were recorded, saliva and GCF samples were obtained before and at first and third months after periodontal therapy. Levels of YKL-40 and IL-6 in saliva and GCF were analyzed by enzyme-linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

Group 1 Inclusion Criteria:

* No bone and attachment loss,
* GI=0, PPD≤3mm, CAL≤3mm
* Systematically healthy patients

Group 2 Inclusion Criteria:

* GI>1, PPD≥5mm, CAL≥5mm with alveolar bone loss radiographically.
* Systematically healthy patients

Exclusion Criteria:

* Aggressive Periodontitis,
* Patients with any other systemic diseases,
* Pregnant women and those in the lactation period,
* Patients with smoking habit and taking medication
* Patients received periodontal therapy in last 6 month

Ages: 26 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 52 participants
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
YKL-40 levels | at first and third month after therapy
  changes in YKL-40 levels after periodontal therapy

SECONDARY OUTCOMES:
IL-6 levels | at first and third month after therapy
  changes in IL-6 levels after periodontal therapy